CLINICAL TRIAL: NCT02935049
Title: Evaluation of the Resection of Adenoma and Colic Adenocarcinoma by EMR Piecemeal or EMR/ESD Hybrid Technique
Acronym: HYBRID ESD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: HYBRID ESD-IPC 2016-015
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Adenoma; Intramucinous Adenocarcinoma
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic resection — Endoscopic resection with technique EMR piecemeal or hybrid technique EMR/ESD

SUMMARY:
For tough colic resection, evaluation of our practice for these lesions unresectable in monoblock and evaluation of the contribution of the hybrid technique EMR (mucosectomy dissection) /ESD (submucosal dissection)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Patient with colorectal adenoma or intramucinous adenocarcinoma

Exclusion Criteria:

* Contraindication surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal adenoma or intramucinous adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | From surgery to 1 year
  Medical follow-up

SECONDARY OUTCOMES:
Complications rate | From surgery to 6 months
  haemorrhage or perforation

CONTACTS AND LOCATIONS:
Overall Officials: RATONE Jean Philippe, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- GENRE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut Paoli-Calmettes — http://www.institutpaolicalmettes.fr